CLINICAL TRIAL: NCT02044757
Title: The Potentially Addictive Properties of Soda: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-08545; 6030sc (Other Grant/Funding Number: UC Office of the President)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Withdrawal Symptoms
Keywords: Caffeine; Addiction; Withdrawal symptoms; Pediatric; Adolescent; Overweight
MeSH Terms: conditions — Substance Withdrawal Syndrome; Behavior, Addictive; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SSB withdrawal (Experimental)
  Interventions: Behavioral: SSB withdrawal

INTERVENTIONS:
Behavioral: SSB withdrawal — During days 1-5, participants will drink the beverages they normally consume (no intervention). On days 6-8, participants will be instructed to drink only water and unflavored milk during the withdrawal period (days 6-8).

SUMMARY:
The purpose of this study to investigate the addictive properties of soda and other sugar sweetened beverages (SBBs) in teenagers aged 13-18 years. It is hypothesized that participants who were regularly consuming sweetened and caffeinated beverages will experience symptoms typical of caffeine withdrawal, such as headache and fatigue, during the SSB withdrawal period.

ELIGIBILITY:
Inclusion Criteria:

* Drinks more than 36 ounces of sugar-sweetened beverages per day
* Speaks fluent English
* Parent speaks English or Spanish
* Lives in San Francisco Bay Area

Exclusion Criteria:

* Pregnant or nursing
* Taking medication to address mental health issues

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Symptoms of withdrawal | Days 1-3 and days 6-8
  Symptoms of withdrawal during the SSB withdrawal period (days 6-8) will be compared to symptoms of withdrawal during usual consumption period (days 1-3). Three measures are used to assess withdrawal symptoms: Griffiths' withdrawal scale, the relative reinforcing value of soda, and daily check in questions on well-being.

SECONDARY OUTCOMES:
Change in diet | Days 1-2, 6-8
  Changes in diet will be assessed by 24-hour dietary recalls and beverage recalls
Change in impulsivity | Days 1 and 8
  Impulsivity will be assessed via the delayed discounting task
Change in stress | Days 1 and 8
  Stress will be assessed via salivary cortisol samples
Change in preference for soda | Days 1-3, 6-8
  Preference for soda will be measured through the Labeled Affective Magnitude Scale (LAMS) and daily check-in questions

OTHER OUTCOMES:
Compliance with intervention to only drink water and unflavored milk during the SSB withdrawal phase | Days 6-8
  Using measure of salivary caffeine, beverage recalls, and 24-hour dietary recalls, we will assess compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD, MPH, Principal Investigator — University of California, Berkeley School of Public Health
Locations (1):
- Children's Hospital and Reasearch Center Oakland, Oakland, California, United States